CLINICAL TRIAL: NCT03469011
Title: A Phase I Dose Escalation Trial to Determine if Imatinib Treatment Restores Sodium Iodide Symporter Function and Sensitivity to Radioiodine Treatment in Metastatic Thyroid Cancer Patients
Brief Title: A Study to Try to Bring Back Radioiodine Sensitivity in Patients With Advanced Thyroid Cancer.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Imatinib-CCI-PH1-01
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imatinib oral100mg tablets (Experimental): A standard 3+3 trial design will be utilized for the imatinib dosing. In general, patients will be treated in cohorts of 3-6 with escalating doses of imatinib using oral 100mg tablets.
  Dose Level -1=100mg, +1=200mg (starting dose for cohort 1), +2=300mg, +3=400mg, +4=600mg (if needed).
  Interventions: Drug: Imatinib Oral Tablet

INTERVENTIONS:
Drug: Imatinib Oral Tablet — 3+3 trial design. Cohorts of 3-6 patients with escalating imatinib doses. No intra-patient dose escalation allowed.
  Other Names: Gleevec

SUMMARY:
Thyroid cancers that have spread beyond the neck are not curable. About 30,000 people worldwide die from thyroid cancer every year. Usually, thyroid cancers get worse because the cancer cells become more and more abnormal through a process that is called dedifferentiation.

Radioactive iodine is a standard treatment for this type of thyroid cancer. Patients will usually receive multiple dose of radioactive iodine over the course of their cancer journey. Thyroid cancers lose sensitivity to radioactive iodine as the cancer progresses/worsens with the process of dedifferentiation. When this occurs, the radioactive iodine treatments no longer work against the cancer and the cancer grows.

Radioactive iodine enters cancer cells through transporter proteins on the outside of the cancer cell. The transporter proteins that are the most important are the sodium iodide symporters. As thyroid cancers dedifferentiate, these symporters stop working as well as they once did. The radioactive iodine can therefore not get into the cancer cells to cause cancer cell death.

Laboratory research has shown that in thyroid cancer, a protein on the cell called platelet derived growth factor receptor alpha (PDGFRα) is an important for tumour growth and thyroid cancer dedifferentiation. PDGFRα helps cancer progression and lowers the ability of sodium iodine symporters to move radioiodine into cells where it would normal act to kill the cancer cells. PDGFRα therefore makes thyroid cells resistant to radioactive iodine.

Imatinib is an anti-cancer drug that blocks PDGFRα function. It has been used for many years to treat other cancers such as leukemia. The investigators who wrote this study believe that, base on laboratory testing, if thyroid cancer patients are given imatinib whenafter their cancers have become resistant to radioactive iodine, the imatinib will block PDGFRα. This will let the sodium iodine symporters work again and move the radioactive iodine into the cancer cells. This should shrink the tumours. Imatinib would then make the thyroid cancer cell sensitive to radioactive iodine again. This should shrink the tumours and would mean longer control of the cancer, helping people with this disease live longer.

DETAILED DESCRIPTION:
This proposed new method of therapy for patients with progressive, metastatic papillary or follicular thyroid cancers will combine a focused blockade of PDGFRα with radioactive iodine. This is based on a new model for dedifferentiation in thyroid cancer as recently published by Lopez-Campistrous et al., 2016 (Appendix 1). Using this model and extensive preclinical data, the investigators hypothesize that the relatively short course of the well-known drug imatinib will allow for re-differentiation of thyroid cancers permitting radioactive iodine transport thus restoring sensitivity to radioactive iodine. The efficacy of these agents will be determined in a trial of 18 patients through a short treatment phase of approximately 3 months through which the investigators should be able to determine a clinically relevant response. The investigators believe this trial is highly clinically relevant and has the benefits of using previously well described treatments in a novel pattern that should maximize efficacy while minimizing toxicity. If successful, this trial will translate into a new treatment paradigm for metastatic thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Cytologically or histologically confirmed papillary thyroid cancer consisting of papillary or follicular variants.

  2. Radioiodine-refractory disease (iodine-refractory thyroid cancer) by at least one of the following criteria:
  1. an index metastatic lesion that was not radioiodine-avid on diagnostic radioiodine scanning performed within 28 days of enrolment;
  2. a radioiodine-avid metastatic lesion that remained stable in size or progressed despite radioiodine treatment 3 months or more before entry into the study; or
  3. 18F-fluorodeoxyglucose (FDG)-avid lesions on PET scan (if available). 3. Recurrent, advanced, or metastatic (Stage IV) disease that is not amenable to surgical resection or radiation with curative intent.

     4. Minimal or no radioactive iodine uptake demonstrated by whole body iodine scans.

     5. Age ≥ 18. 6. Eastern Cooperative Oncology (ECOG) performance status of ≤ 1. 7. Presence of measurable disease, defined as at least 1 unidimensional measurable lesion on a computed tomography (CT) scan as defined by RECIST 1.1.

     8. Hematology: WBC ≥ 3.0 x 109/L or granulocytes (polymorphs + bands) ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L within 4 weeks prior to enrolment.

     9. AST (SGOT) and/or ALT (SGPT) and alkaline phosphatase ≤ 5 x the upper limit of normal (ULN). Creatinine ≤ 1.5 x ULN.

     10. Serum amylase and lipase ≤ 1.5 x ULN 11. Serum potassium, phosphorus, magnesium and calcium ≥ lower limit of normal or correctable with supplements prior to first dose of study drug.

     12. Be able to comply with study procedures and follow-up examinations. 13. Not pregnant or lactating. Male and female patients who are fertile must agree to use an effective means of birth control (i.e., latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy.

     14. Sign a written informed consent.

     Exclusion Criteria:
* 1. Has received radiation therapy within 21 days of Study Day 1. 2. Has had major surgery within 21 days of Study Day 1. 3. Has untreated brain or meningeal metastases. Patients who have treated brain metastasis (via local radiation standards or surgical resection or local ablative techniques) and who are either off steroids or on a stable dose of steroids for at least one month (30 days), AND who are off anticonvulsants, AND have radiological documented stability of lesions for at least 3 months may be eligible. Each case should be discussed with the Principal Investigator.

  4. Has a central thoracic tumor lesion as defined by location within the hilar structures.

  5. Has proteinuria CTCAE v.4.0 Grade > 1 at baseline. 6. Has a history of, or currently exhibits clinically significant cancer related events of bleeding.

  7. Currently exhibits untreated, symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure (BP) > 90 mm Hg or systolic BP > 140 mm Hg.

  8. Has a history of myocardial infarction, stroke or Transient Ischemic Attack (TIA) within 6 months of Study Day 1.

  9. Impaired cardiac function including any of the following:
  1. Has a documented left ventricular (LV) ejection fraction < 50%;
  2. Long QT syndrome or family history of long QT syndrome;
  3. Clinically significant resting bradycardia (<50 bpm);
  4. Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, unstable angina, significant ventricular or atrial tachyarrhythmia).

     10. Treatment with strong CYP3A4 inhibitors (e.g. erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.

     11. Treatment with strong CYP3A4 inducers (e.g. dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's Wort), and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.

     12. Patients using medication that have been documented to prolong QT interval should be avoided. In the case it is not possible to avoid or switch to other medication, patients should be followed with caution and ECG testing should be requested at least every 3 months after starting study or if any dose change occurs or if clinical symptoms appear.

     13. Has known autoimmune disease with renal involvement (e.g. lupus). 14. Receiving combination anti-retroviral therapy for HIV. 15. Has clinically significant uncontrolled condition(s). 16. Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or uterus or non-melanoma skin cancer or in-situ carcinoma of the prostate (Gleason score ≤ 7, with all treatment being completed 6 months prior to enrollment, unless at least 5 years have elapsed since last treatment and the patient is considered cured).

     17. Has active ulcerative colitis, Crohn's disease, celiac disease, short gut syndrome from any cause, or any other conditions that interfere with absorption.

     18. History of acute pancreatitis within one year of study entry or medical history of chronic pancreatitis.

     19. Has a medical condition, which in the opinion of the study investigator places them at an unacceptably high risk for toxicities.

     20. Pregnant or breast feeding. 21. History of non-compliance to medical regimens or inability to grant consent.

     22. Use of an investigational agent within 28 days prior to enrollment in the study or foreseen use of an investigational agent during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Restore iodine uptake | 3 months
  To demonstrate that imatinib can restore iodine uptake in iodine-refractory thyroid carcinoma, as determined by whole body iodine scans.

SECONDARY OUTCOMES:
Decrease overall tumor burden | 3 months
  To determine if treatment with imatinib and radioactive iodine ablation can decrease overall tumor burden through restored sodium iodide symporter function in iodine-refractory thyroid carcinoma. This will be assessed by thyroglobulin levels and by anatomic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Todd McMullen, Principal Investigator — Alberta Health services; Jennifer Spratlin, MD FRCPC, Principal Investigator — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No